CLINICAL TRIAL: NCT04075942
Title: Horizontal Ridge Reconstruction of Atrophic Anterior Maxillary Ridges Using Customized Xenograft Bone Shell With 1 :1 Mixture of Autogenous and Xenograft Bone Particulate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Manal Ahmed Hassan Ahmed (Other)
Responsible Party: Sponsor-Investigator, Manal Ahmed Hassan Ahmed, Faculty of dentistry, Master degree of dental Implantology, Cairo University
Organization: Cairo University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PER 6-3-1
Record Dates: First submitted 2019-08-28; First posted 2019-09-03 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Atrophic Anterior Maxillary Ridges

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atrophic Anterior Maxillary Ridges participants (Other): Using customized Xenograft bone shell with equal mixture of autogenous and xenograft particulate bone as a graft with the modified cortical shell technique, with atrophic anterior maxilla with less than 5 mm Bucco-lingual
  Interventions: Procedure: Atrophic Anterior Maxillary Ridges

INTERVENTIONS:
Procedure: Atrophic Anterior Maxillary Ridges — Use of modified cortical shell technique grafted with customized Xenograft bone shell

SUMMARY:
Using customized Xenograft bone shell with mixture of autogenous and xenograft particulate in modified cortical shell technique. by 3D printed model from The CT scans segmentation by special software

DETAILED DESCRIPTION:
Using customized Xenograft bone shell by 3D printed model from The CT scans segmentation by special software ( Mimics ) . All surgeries were performed by the same surgeon .

All surgical procedures were performed under strict aseptic conditions, all patients received infiltration local anesthesia (Articaine 4% 1:100 000 epinephrine).

a midcrestal incision was made in the anterior region using No. 15 blade. A full thickness mucoperiosteal flap was raised to expose the underlying alveolar ridge. The residual remaining bone in the area was minimal, with a maximum measured ridge thickness of 3 or 4 mm. 'To reconstruct the lost alveolar bone, an xenograft bone shell approximately 1 to 2 mm thick was shaped, after 3D print the bone shell were fixed to the buccal defect, using screws . 'The space between the plate and the existing palatal bone wall was then filled using a combination of autograft bone chips and xenograft bone particles

. Periosteal releasing incision is done to obtain stress free primary closure. The flap will then be closed using interrupted 4/0 resorbable sutures. After 4 month will insert implant . After 3 month will insert final restoration which will be mostly PMF .

ELIGIBILITY:
Inclusion Criteria:

* patients with atrophic Anterior Maxillary Ridges

Exclusion Criteria:

* Heavy smokers
* Uncontrolled diabetic patients.
* Pregnant patients. Psychiatric patient
* pathology related to bone.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Bucco-lingual bone width gain. | 4 months

IPD SHARING:
Plan to Share IPD: No